CLINICAL TRIAL: NCT05177718
Title: Assessing the Effect of Natalizumab of Magnetic Resonance Imaging Measures of Blood Brain Barrier Permeability and Myelin Integrity
Brief Title: Natalizumab and Chronic Inflammation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor declined further support
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Francesca Bagnato, Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201600
Record Dates: First submitted 2021-12-13; First posted 2022-01-05 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis, MRI, blood brain barrier, myelin
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab; Injections

STUDY DESIGN:
Intervention Model Description: Open-label, prospective longitudinal study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Single Arm (Other): SINGLE ARM: 30 patients with multiple sclerosis treated with Natlizumab infusion given monthly at the dose of 300 mg IV
  Interventions: Drug: Natalizumab 300 MG in 15 ML Injection

INTERVENTIONS:
Drug: Natalizumab 300 MG in 15 ML Injection — Disease modifying agent

SUMMARY:
In this study the investigators will assess the ability of Natalizumab, a medication given to treat multiple sclerosis (MS), to restore blood brain barrier integrity and repair subtle leakages of the blood brain barrier (BBB).

DETAILED DESCRIPTION:
The investigators will image a cohort of persons with relapsing remitting multiple sclerosis (pwRRMS) using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) and selective inversion recovery quantitative magnetization transfer imaging (SIR-qMT). pwRRMS will be imaged at baseline and at month-3 and month-12, after starting treatment with natalizumab. Changes in ktrans, a measure of BBB permeability derived from DCE-MRI, and in pool saturation ratio (PSR) a measure of myelin integrity derived from SIR-qMT will be computed to assess the ability of natalizumab to fully restore BBB integrity.

As a corollary aim, the investigators will assess changes in quality of life (QoL) measurements and the relation between those measurements and those derived from the above detailed quantitative MRI methods. QoL will be measured using the Visual Analogue Scale. This questionnaire entails 13 questions regarding the perceived effect of Tysabri, but also level of pain, fatigue, anxiety, depression before and during treatment with natalizumab. The answer to each question is rated on a color-coded bar the range of which is between 0 to 100.

ELIGIBILITY:
Inclusion Criteria:

1. multiple sclerosis
2. clinical eligibility to treatment with Natalizumab
3. no previous exposure to Natalizumab treatment

Exclusion Criteria:

1. inability to perform an MRI with contrast
2. inability to undergo a paper-pencil questionnaires and blood work

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Bagnato, MDPhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request from qualified investigators the PI will release all data listed below.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: [per PDBP policy]
Access Criteria: [per PDBP policy]
URL: https://pdbp.ninds.nih.gov/policy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Single Arm
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Single Arm
Number analyzed (Participants) | 1
Age, Customized [Number; unit: years]
  46 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Effect of Natalizumab on Magnetic Resonance Imaging Measures of Blood Brain Barrier Permeability: K-trans
Description: To measure changes in k-trans between baseline (pre-treatment) and month-3 and month-12 post-treatment scan
Time Frame: 12 months
Population: Data analysis was not completed because only one participant completed (each arm) and disclosing data could violate privacy interests.
Groups:
- Single Arm: Treatment with natalizumab at standard dose
Arm/Group | Single Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Effect of Natalizumab on Magnetic Resonance Imaging Measures of Myelin Integrity: Pool Saturation Ratio (PSR)
Description: To measure changes in PSR between baseline (pre-treatment) and month-3 and month-12 post-treatment scan
Time Frame: 12 months
Population: Data analysis is not reported because only one participant completed (each arm) and disclosing data could violate privacy interests.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Effect of Natalizumab on Questionnaire Derived Measures of Quality of Life
Description: To explore changes in QoL measurements and the relations between these changes and those seen in ktrans and natalizumab serum levels.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: At baseline, month 3 and month 12.
Description: Adverse events were collected and reviewed by the PI
Arm/Group | Treatment Single Arm
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT05177718/Prot_SAP_000.pdf